CLINICAL TRIAL: NCT04403724
Title: Comparison of Sequential and Mixture Injection of Opioids and Hyperbaric Bupivacaine for Subarachnoid Block for Elective Caesarean Section; a Randomised Controlled Study
Brief Title: Sequential and Mixture Injection of Opioids and Hyperbaric Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300377 (sequential)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Bupivacaine Adverse Reaction; Regional Anesthesia Morbidity; Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- premixed injection (Active Comparator): will receive an intrathecal injection of 2.4 ml hyperbaric bupivacaine 0.5%, 20 µg fentanyl, and 100 µg preservative-free morphine mixed together.
  Interventions: Drug: Bupivacaine-fentanyl-Morphine.
- sequential injections (Active Comparator): will receive an intrathecal injection of 2,4 ml hyperbaric bupivacaine 0.5% followed immediately by the opioid mixture by two separate syringes.
  Interventions: Drug: Bupivacaine-fentanyl-Morphine.

INTERVENTIONS:
Drug: Bupivacaine-fentanyl-Morphine. — 2.4 ml Bupivacaine 0.5%, 20 µg Fentanyl and, 100 µg preservative free morphine

SUMMARY:
Neuraxial anesthesia, especially the subarachnoid block, is the preferred method for LSCS. The intrathecal spread of local anesthetic drugs is unpredictable. However, Baricity, which is the relative density of local anesthetics to that of CSF, is a key determinant of the local anesthetic spread within the subarachnoid space. Alterations in the baricity of a solution to the extent of 0.0006 g/ml-1 can alter the spread of local anesthetic solution in CSF. Patients features such as position, weight, height, and age, and local anaesthetic characteristics such as density, PH, and temperature may play a role as well.

Bupivacaine is the main local anaesthetic used frequently for the subarachnoid block. Hyperbaric bupivacaine has dextrose added at a concentration of 80 g/ml to increase its density to 1.0262 which is higher than that of cerebrospinal fluid (CSF), leading to a more predictable spread after intrathecal injection.

Opioids such as morphine and fentanyl are commonly injected as adjuvants to hyperbaric bupivacaine. Their synergistic role leads to satisfactory block at smaller subtherapeutic doses of bupivacaine which minimizes the associated side effects. The combination of fentanyl which is lipophilic opioid and morphine which is hydrophilic opioid results in rapid onset and prolonged course of perioperative analgesia. In an in vitro study, the mean densities of fentanyl and morphine were found to be 0.9957 and 1.0013 respectively while the mean density of CSF in term pregnant woman is 1.000306. Thus, opioids spread freely within the CSF interacting on the spinal and supraspinal opioid receptors. They have a synergistic effect to bupivacaine leading to adequate sensory blockade with lesser hemodynamic adverse effects.

Nevertheless, opioids are commonly mixed with hyperbaric bupivacaine in a single syringe before intrathecal injection. This practice alters the density and PH of the mixture which may impact the pharmacokinetics of each individual drug. Therefore, we hypothesize in this study that separate injection of opioids and hyperbaric bupivacaine may improve their intrathecal spread. This will not only improve the quality of anesthesia, but it will also decrease the associated hemodynamic adverse events and the incidence of undesired high sensory block levels, which all will increase the perioperative patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* LSCS
* ASA I or II
* Single baby pregnancy of more than 32 weeks
* Elective or semi-elective surgery (category 3 and 4 Caesarean sections)

Exclusion Criteria:

* Abnormal Placentation
* PET
* Disordered coagulation
* Allergy to opioids or local anesthetic.
* BMI > 35
* Spine surgery
* Cardiac disease
* Extremes of height; height more than 180 or less than 140
* Multiple pregnancy or polyhydramnios

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
duration to the maximal sensory block to light touch | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Egypt

REFERENCES:
- [Derived] Moustafa MMI, Ali MS, McCaul C, Abbas MS. Comparison of sequential and mixture injections of opioids and hyperbaric bupivacaine for subarachnoid block for lower segment caesarean section: a randomised controlled study. Ir J Med Sci. 2024 Aug;193(4):1977-1983. doi: 10.1007/s11845-024-03682-w. Epub 2024 Apr 11. PMID 38602618